CLINICAL TRIAL: NCT03030885
Title: A Phase 1, Open-Label, Dose Ascending Study to Evaluate the Safety and Tolerability of the Therapeutic Radiopharmaceutical 131I-MIP-1095 for the Treatment of Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Use of an Experimental Radiopharmaceutical (131I-MIP-1095) in Men With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1110
Record Dates: First submitted 2017-01-22; First posted 2017-01-25 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer; Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Radiopharmaceutical (131I-MIP-1095); 16-1110
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label, single-arm, dose ascending, out-patient study to evaluate the radiopharmaceutical 131I-MIP-1095 in men with mCRPC. The study consists of three phases: Screening, Treatment, and a Follow-up Phase. The Screening Phase consists of subject evaluation for study eligibility and dosimetry assessment. The Treatment Phase consists of two parts: Part 1, dose escalation (Cohorts 1-5), and Part 2, an additional cohort at a selected optimized dose based on safety and efficacy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 131I-MIP-1095 (Experimental): FirstTherapeutic Dose with 131I-MIP-1095 to be administered no later than 30 days after dosimetry dose, which will be designated Day 1 of the Treatment Phase 2nd and 3rd Therapeutic Doses with 131I-MIP-1095 to be administered 12 weeks apart Monthly Follow-Up Visits until Week 41. 1st Therapeutic Dose with 131I-MIP-1095 to start after qualifying from dosimetry on Day 8 or no later than 30 days after dosimetry dose.
  2nd and 3rd Therapeutic Doses with 131I-MIP-1095 to be administered 12 weeks apart Monthly Follow-Up Visits until Week 53
  Interventions: Drug: 131I-MIP-1095

INTERVENTIONS:
Drug: 131I-MIP-1095 — First Therapeutic Dose with 131I-MIP-1095 to be administered no later than 30 days after dosimetry dose, which will be designated Day 1 of the Treatment Phase 2nd and 3rd Therapeutic Doses with 131I-MIP-1095 to be administered 12 weeks apart Monthly Follow-Up Visits until Week 41. 1st Therapeutic Dose with 131I-MIP-1095 to start after qualifying from dosimetry on Day 8 or no later than 30 days after dosimetry dose.
  2nd and 3rd Therapeutic Doses with 131I-MIP-1095 to be administered 12 weeks apart Monthly Follow-Up Visits until Week 53

SUMMARY:
The main purpose of this study to determine the safety of an experimental medicine called 131I-MIP-1095. 131I-MIP-1095 is an investigational drug, meaning it has not been approved by the U.S. Food & Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Males, age ≥18 years.
* Subjects must have histologically or cytologically confirmed adenocarcinoma of the prostate
* Subjects must be castration resistant with evidence of progressive prostate cancer despite castrate levels of testosterone (≤ 50 ng/dL) according to the PCWG3 criteria
* Subjects must have metastatic disease detectable by either bone scan or cross sectional imaging by CT or MRI as per the PCWG3 guidelines
* Subjects must have progressive disease at study entry defined as 1 or more of the following 3 criteria that occurred while the subject was on androgen deprivation therapy:

  * PSA progression defined by a minimum of two rising PSA levels with an interval of ≥1 week between each determination. Subjects who received an anti-androgen as part of their primary hormonal therapy must demonstrate progression after withdrawal. The PSA value at screening should be ≥ 2 μg/L (2 ng/mL).
  * Soft tissue disease progression defined by RECIST 1.1
  * Bone disease progression defined by PCWG3 with two or more new lesions on bone scan.

Note: For subjects enrolling on the basis of soft tissue or bone progression, the baseline scan must show progression relative to a comparison scan performed during prior therapy. If the comparison scan is not available, the baseline scan report must reference the previous scan to document progression

* Subjects who received combined androgen blockade as their first-line hormonal therapy with an antiandrogen must have shown PSA progression after discontinuing the antiandrogen for ≥ 6 weeks prior to study treatment. No washout is needed after abiraterone or enzalutamide are discontinued. First generation antiandrogens such as bicalutamide must be withdrawn if given as first-line therapy.
* ECOG Performance status of 0-1.
* Adequate organ reserve as evidenced by:

  1. neutrophil count ≥ 1500 μL
  2. platelet count ≥ 100,000/μL
  3. hemoglobin ≥ 9.5 g/dL
  4. total bilirubin level ≤1.5 x ULN
  5. AST and ALT ≤2.5 x ULN
  6. serum amylase ≤ ULN
  7. lipase ≤ ULN
  8. serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥ 60 mL/min (Cockroft Gault equation)
  9. clearance of 99mTc MAG3 within 1.5 x ULN and no evidence of obstruction on the scan.
* Serum albumin of > 3.0 g/dL
* Subjects must have received, were ineligible to receive, or refused at least one cytotoxic chemotherapy and enzalutamide or abiraterone or both enzalutamide and abiraterone.
* Subjects must agree to use a medically acceptable method of birth control (e.g., spermicide in conjunction with a barrier such as a condom) or sexual abstinence for the duration of the study, including 30 days after the last dose of study drug. Sperm donation is prohibited during the study and for 30 days after the last dose of study drug. Female partners must use hormonal or barrier contraception unless postmenopausal or abstinent.
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Subject has predominant histologically or cytologically confirmed neuroendocrine prostate cancer (mixed histology is permissible, as is positivity of serum CgA and CEA).
* Subject has received an investigational therapeutic agent for prostate cancer within 4 weeks prior to the administration of 131I-MIP-1095.
* Subject who has not recovered from the effects of any major surgery prior to initial treatment
* Subject has received treatment with a systemic therapeutic radioisotope (89Sr, 223Ra dichloride, 153Sm-lexidronam) or has received prior external beam radiation therapy (EBRT) of the head and/or neck.
* Subject is currently on renal dialysis
* Subject has started treatment with denosumab < 1 month prior to study entry. Subjects are allowed to be on bisphosphonates or denosumab provided they are on a stable dose for ≥ 4 weeks before administration of study drug
* Subject using chronic systemic steroids greater than the equivalent of 10 mg of prednisone/prednisolone per day in the 2 weeks preceding study entry ; replacement doses of steroids, topical, inhalational, nasal and ophthalmic steroids are permitted.
* Diagnosis of other invasive malignancies within the preceding 3 years prior to screening with > 30% likelihood of relapse within the next 3 years, except non-melanoma skin cancer and non-muscle invasive urothelial cancer
* Any other serious illness or medical condition or social circumstance that might interfere with the subject's participation in the trial or interfere with the interpretation of the results, including, but not limited to:

  1. any uncontrolled infection
  2. NYHA Class III or Class IV heart failure
  3. unstable angina
  4. myocardial infarction within the 6 months prior to study entry
  5. uncontrolled hypertension (systolic BP > 160 mmHg despite 2 antihypertensive medications)
  6. COPD requiring hospital admission in the year prior to study entry
  7. diabetes mellitus requiring hospital admission in the year prior to study entry
  8. chronic liver disease
  9. hypothyroidism (TSH level > 3.0 mIU/L)
  10. substance abuse
* Unable or unwilling to follow post-therapy radiation protection procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 years
  This is a phase 1 dose escalation study of 131I-MIP-1095 in men with metastatic castration-resistant prostate cancer. There are a maximum of five doses under consideration. Dose escalation cohorts will be studied if acceptable toxicity is observed. A dose limiting toxicity is defined as the occurrence of any of the following drug-related toxicities during the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Laccetti AL, Bodei L, O'Donoghue JA, Weber WA, Morris MJ. A Phase 1, Open-label, Dose-Ascending Study to Evaluate the Safety and Tolerability of the Therapeutic Radiopharmaceutical 131I-MIP-1095 for the Treatment of Metastatic Castration-Resistant Prostate Cancer. Clin Nucl Med. 2023 Nov 1;48(11):937-944. doi: 10.1097/RLU.0000000000004818. PMID 37812518
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm